CLINICAL TRIAL: NCT01566058
Title: Pilot Study Evaluating the Impact of the BB Box System on Postpartum Maternal Anxiety, Post Traumatic Stress and the Establishment of a Mother-child Relationship in the Context of a Premature Birth
Brief Title: Impact of the BB Box System on Postpartum Maternal Anxiety, Post Traumatic Stress and Mother-child Relationships
Acronym: BBBox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2011/FBC-01; 2012-A00327-36 (Other: RCB number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Stress Disorders, Post-Traumatic; Anxiety
Keywords: Post partum; mother-child relationships
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With BB Box (Experimental): The mothers in this arm of the study will have access to a "BB Box" video system to maintain contact with their premature baby.
  Interventions: Device: BB Box available
- Without BB Box (Active Comparator): The mothers in this arm of the study will not have access to a "BB Box" video system to maintain contact with their premature baby. (Standard care)
  Interventions: Other: No BB Box

INTERVENTIONS:
Device: BB Box available — The BB Box video system is provided to the mother during the hospitalisation of her premature baby.
  Arms: With BB Box
Other: No BB Box — The BB Box video system is not provided to the mother during the hospitalisation of her premature baby.
  Other Names: Standard care
  Arms: Without BB Box

SUMMARY:
The main objective of this study is to compare the degree of maternal anxiety at Day 3 postpartum in mothers who did or did not have access to a video communication system (BB-Box system) from the time of initial separation with their baby.

DETAILED DESCRIPTION:
The secondary objectives of the study are to compare the following between the two arms of the study:

A. The degree of postpartum maternal anxiety at day 1, day 7 and at hospital discharge. Anxiety will be compared point by point but also via kinetics.

B. The incidence maternal post traumatic stress disorder at 6 and 12 months.

C. The incidence of mother-child relationship disorders at 6 and 12 months.

D. Infant vital signs during the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 12 months of follow up
* The patient has given birth this day to a premature child (< 36 weeks of gestation and/or < 2 kg birthweight)
* Separation of child and mother since birth

Exclusion Criteria:

* The patient or baby is participating in another study, excepting the studies "OASIS" or "PROM8736"
* The patient or baby is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient or father refuses to sign the consent
* It is impossible to correctly inform the patient
* Preexisting maternal psychiatric pathology
* Major or lethal poly-malformation syndrome
* Severe pathologies that threaten child survival: pulmonary hypertension, septic shock, anoxic-ischemic brain
* Any emergency situation preventing patient involvement
* Mother and/or child not hospitalized at the Nîmes University Hospital
* Death of the patient or child during the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Questionnaire HADS | Day 3 post-partum
  Score ranging from 0 - 21

SECONDARY OUTCOMES:
Questionnaire HADS | baseline; day 0
  score ranging from 0 to 21
Questionnaire HADS | Day 1 post partum
  score ranging from 0 to 21
Questionnaire HADS | Day 7 post partum
  score ranging from 0 to 21
Questionnaire HADS | Day of hospital discharge for the baby (expected average of 4 weeks)
  score ranging from 0 to 21
Questionnaire PPQ (post traumatic stress disorder) | 6 months post partum
  score ranging from 0 to 14
Questionnaire PPQ (post traumatic stress disorder) | 12 months post partum
  score ranging from 0 to 14
Massie Campbell scale for mother-child relationships | Day of hospital discharge for the baby (expected average of 4 weeks)
Massie Campbell scale for mother-child relationships | 6 months post partum
Massie Campbell scale for mother-child relationships | 12 months post partum
Number of infant cardiovascular events | base line to day of hospital discharge for the baby (expected average of 4 weeks)
  includes bradycardia < 100/min and O2 saturation < 60%

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Benito-Castro, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France